CLINICAL TRIAL: NCT05492110
Title: REducing Microvascular Dysfunction in Patients With Angina, Ischaemia and unobstructED coronarY Arteries - a PILOT Study
Brief Title: Coronary Sinus Reducer Implantation in Patients With Ischaemia and Non-obstructed Coronary Arteries and Coronary Microvascular Dysfunction.
Acronym: REMEDY-PILOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Bradford Teaching Hospitals NHS Foundation Trust (Other Government); East and North Hertfordshire NHS Trust (Other Government); Epsom and St Helier University Hospitals NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); Kingston Hospital NHS Trust (Other); London North West Healthcare NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21IC7301
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Refractory Angina; Microvascular Angina; Microvascular Coronary Artery Disease; Coronary Disease; Angina Pectoris
Keywords: Angina pectoris; Refractory angina; Microvascular angina; Coronary microvascular dysfunction; Coronary sinus reducer; Chest pain; Coronary disease; Myocardial ischaemia
MeSH Terms: conditions — Angina Pectoris; Microvascular Angina; Coronary Disease; Chest Pain; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomised, double-blinded, sham-controlled pilot study with parallel arms of participants randomised to CS Reducer or sham procedure
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be randomised and blinded to CS Reducer of sham procedure. All follow-up assessments will be performed by a blinded parallel team to ensure blinded outcomes analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CS Reducer implantation (Active Comparator)
  Interventions: Device: Coronary sinus reducer; Diagnostic Test: Invasive coronary physiology
- Sham procedure (Sham Comparator)
  Interventions: Other: Sham-procedure; Diagnostic Test: Invasive coronary physiology

INTERVENTIONS:
Device: Coronary sinus reducer — The Neovasc coronary sinus reducer is an hourglass-shaped stainless steel device inserted percutaneously into the coronary sinus and currently indicated for the treatment of refractory angina.
  Arms: CS Reducer implantation
Other: Sham-procedure — Implantation procedure with no device implanted
  Arms: Sham procedure
Diagnostic Test: Invasive coronary physiology — Invasive coronary physiology assessment as part of REMEDY-MECH mechanistic substudy

SUMMARY:
To demonstrate the feasibility and efficacy of the CS Reducer for the treatment of patients with ischaemia and non-obstructed coronary arteries (INOCA) and coronary microvascular dysfunction (CMD) and through a nested mechanistic substudy investigate the physiological responses in the coronary microcirculation responsible for changes in myocardial perfusion.

DETAILED DESCRIPTION:
Symptomatic angina in patients with ischaemia and non-obstructed coronary arteries (INOCA) is common and associated with increased morbidity and adverse outcomes. Myocardial ischaemia often arises from coronary microvascular dysfunction (CMD). Current treatments are limited, and novel evidence-based therapies are needed to address this large unmet clinical need. The Coronary Sinus Reducer (CS Reducer) is a new treatment for refractory angina, which creates a focal narrowing in the coronary sinus that increases back pressure and redistributes blood into ischaemic myocardium at the level of the microcirculation. However the precise mechanism remains unknown. This study will be a randomised double-blinded sham-controlled pilot study (REMEDY-PILOT) to confirm acceptability of CS Reducer implantation, demonstrate feasibility to recruit and quantify its effect on myocardial perfusion. A nested mechanistic substudy within REMEDY-PILOT will test the hypothesis that CS Reducer implantation alters measures of invasive coronary microcirculatory physiology as the mechanistic basis for observed changes in quantitative CMR stress perfusion, symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Ongoing symptomatic angina, CCS Class II-IV, for ≥3 months despite background treatment with at least two anti-anginal drug at the maximal tolerated dose.
3. Patients willing to consider no change in anti-anginal drug treatment for the duration of their participation in the trial.
4. Unobstructed coronary arteries with ≤50% epicardial stenoses demonstrated on coronary angiography.
5. Stress-induced hypoperfusion on CMR (Global MPR ≤ 2.2).
6. Willingness to comply with the specified follow-up evaluation and to be contactable during the period of the trial.
7. Understands the nature of the trial procedures and provides written informed consent.

Exclusion Criteria:

1. Epicardial CAD in a main coronary artery (stenoses >50%, RFR≤0.92 or FFR≤0.80), coronary artery bypass grafting, or myocardial infarction (MI).
2. Previous PCI within 6 months
3. PCI with stent insertion for acute MI or chronic total occlusion (CTO)
4. Abnormal coronary sinus anatomy (tortuosity, aberrant branch, persistent left superior vena cava)
5. Coronary sinus diameter at site of implant <9.5mm or >13mm
6. Mean right atrial pressure <15mmHg at time of implantation
7. Any structural heart disease including left ventricular hypertrophy; cardiomyopathy; severe valvular heart disease; previous valve replacement; myocardial bridge on angiography; LVEF<45% by CMR.
8. Clinically or angiographically diagnosed coronary vasospasm
9. Previous hospitalisation for decompensated heart failure
10. Pacemaker or defibrillator electrode in the right atrium, right ventricle or coronary sinus
11. Documented arrhythmia requiring planned implantation of a permanent pacemaker or defibrillator
12. Chronic kidney disease (creatinine >200 micromol/L; established on renal replacement therapy; functioning renal transplant)
13. Haemoglobin <80g/L
14. Contraindications to receiving dual antiplatelet therapy
15. Severe chronic obstructive pulmonary disease (FEV1 <55% predicted)
16. Moribund patients with life expectancy < 1year
17. Known allergy to nickel or steel
18. Current enrolment in another investigational device or drug trial
19. Contraindications to CMR or receiving intravenous adenosine
20. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
number of patients consenting to participate in the study. | 6 months
  Consent rate
Premature withdrawal rate including reasons for withdrawal | 6 months
  Registry of patients either failing screening or unwilling to consent to full trial
Change in myocardial perfusion | 6 months
  Change at 6 months post randomisation, compared to baseline, in quantitative myocardial perfusion (global myocardial perfusion reserve [MPR]) assessed by cardiac MRI.

SECONDARY OUTCOMES:
Canadian Cardiovascular Society (CCS) Angina Score | 6 months
  Change in CCS class from baseline to 6 months post-randomisation. The CCS grading system for angina is a clinical tool used by doctors to assess the degree of severity of a patient's angina. Possible scores range from Class 0 (asymptomatic angina) to Class IV (angina at rest).
Seattle Angina Questionnaire (SAQ) score | 6 months
  Change in SAQ score from baseline to 6 months. The Seattle Angina Questionnaire (SAQ) is a disease-specific questionnaire used to quantify patients' symptoms of angina and the extent to which their angina affects their functioning and quality of life. Possible scores range from 0 (daily angina) to 100 (no angina). Lower scores indicate worse angina symptoms.
Short-form 36 (SF-36) | 6 months
  Change in SF-36 scores from baseline to 6 months. Validated questionnaire to assess quality of life. 36 items each scored from 0-100 with higher scores indicating a more favourable health state.
Hospital Anxiety and Depression Scale (HADS) | 6 months
  Change in HADS score from baseline to 6 months. Scores range from 0 to 21. Normal results are indicated by lower scores. Validated questionnaire to assess psychological wellbeing.
6-minute walk test (6MWT) | 6 months
  Change in exercise capacity from baseline to 6 months. Distance in metres walked in 6 minutes.
BORG scale of perceived exertion | 6 months
  Change in BORG scale from baseline to 6 months. Scores range from 0 to 20 (BORG scale) or 0 to 10 (Modified BORG scale). The higher the self-reported score, the greater perceived exertion.
Safety events - rate of major adverse events | 6 months
  The rate of occurrence of a composite of death, myocardial infarction (MI), pericardial effusion requiring surgical or percutaneous intervention, device embolisation, or BARC 3 or 5 bleeding evaluation in the CS Reducer arm compared to the sham-procedure arm.

OTHER OUTCOMES:
Change in absolute global myocardial perfusion (ml/min/g) at rest and during adenosine stress (transmural, endocardial, epicardial) from baseline to 6 months post-randomisation | 6 months
Change in absolute myocardial perfusion (ml/min/g) at rest and during adenosine stress (transmural, endocardial, epicardial) from baseline to 6 months post-randomisation in the distribution territory of the left coronary circulation. | 6 months
Change in global endocardial:epicardial perfusion ratio at rest and after adenosine stress from baseline to 6 months post-randomisation | 6 months
Change in endocardial:epicardial perfusion ratio at rest and after adenosine stress from baseline to 6 months post-randomisation in the distribution territory of the left coronary circulation. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ranil E de Silva, FRCP, PhD, Principal Investigator — Imperial College London
Locations (1):
- National Heart and Lung Institute (Brompton Campus), Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No